CLINICAL TRIAL: NCT04198337
Title: Prospective Clinical Study on Safety and Effectiveness of Endoscopic Full Thickness Resection for Treatment of Patients With Gastric Gastrointestinal Stromal Tumors (GIST)
Brief Title: Endoscopic Full Thickness Resection for Gastric GIST
Acronym: EFTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC 2014.293-T
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Gastric GIST
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic Full Thickness Resection (Experimental): Resection of the gastric GIST by ESD techniques followed by endoscopic closure of defect with suturing or clips and loop
  Interventions: Procedure: Endoscopic Full Thickness Resection

INTERVENTIONS:
Procedure: Endoscopic Full Thickness Resection — Endoscopic full thickness resection achieved by resecting the submucosal tumor using retraction techniques and submucosal dissection, followed by closure

SUMMARY:
This is a clinical trial to evaluate the efficacy and safety of endoscopic full thickness resection for treatment of gastric GIST

DETAILED DESCRIPTION:
To evaluate the clinical safety and efficacy of endoscopic full thickness resection (EFTR) for treatment of gastric GIST. A total of 30 patients will be recruited

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and ≤ 80
2. Gastric submucosal tumors located at cardia, lesser curvature and antrum
3. Size of the submucosal tumor between 10mm to 30mm as assessed by endoscopic

Exclusion Criteria:

1. Patients who are considered as unfit for general anesthesia
2. ASA class ≥ IV or moribund patients
3. Pregnancy
4. Gastric submucosal tumors located at greater curvature and fundus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete resection of GIST | 30 days
  Complete resection of the GIST defined by en-bloc resection in one piece by endoscopy with clear resection margins

SECONDARY OUTCOMES:
Adverse event rate | 30 days
  Adverse event as defined by presence of either postoperative bleeding or leakage after closure
Perioperative mortality | 30 days
  Death within 30 days after procedure
Histolology assessment | 30 days
  Histology outcome as defined by any involvement of the tumor margins after resection
Hospital stay | 30 days
  Length of stay in hospital
technical success in complete resection | 1 day
  Technical success defined by complete endoscopic resection, closure of the defect and delivery of the specimen per orally without need of conversion to laparoscopic surgery

CONTACTS AND LOCATIONS:
Overall Officials: Philip Wai Yan Chiu, MD, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Outside of US & Canada, China

IPD SHARING:
Plan to Share IPD: Undecided